CLINICAL TRIAL: NCT04240496
Title: Clinical and Genetic Influencing Factors on Clozapine Pharmacokinetics in Schizophrenic Patients
Brief Title: Clinical and Genetic Influencing Factors on Clozapine Pharmacokinetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Dr. Helmi AMMAR, Resident Doctor, University of Monastir
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IORG 0009738 N°30
Record Dates: First submitted 2020-01-16; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: CYP1A2 Polymorphism; CYP2C19 Polymorphism; Clozapine; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Genotype

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Schizophrenic patients (Other): * Determination of trough plasma concentration of clozapine (C0)
  * Genotyping of CYP1A2 & CYP2C19 Drug: Leponex (Clozapine) : was started at a dose of 25 mg/j, the dose was gradually increased and was administered in one, two or three divided doses.
  Interventions: Other: Determination of plasma concentration of clozapine/ Genotyping

INTERVENTIONS:
Other: Determination of plasma concentration of clozapine/ Genotyping — Determination of trough plasma concentration of clozapine (C0) Genotyping of CYP1A2 & CYP2C19

SUMMARY:
Clozapine (Clz), an atypical antipsychotic, is the reference medication for patients with treatment-resistant schizophrenia. Due to the high inter-individual variability of its pharmacokinetics and its narrow therapeutic index, a close therapeutic drug monitoring (TDM) of Clz is highly recommended.

Several factors can cause a variation in the pharmacokinetics as age, smoking habits, coffee consumption and drug interaction. Genetic factors related to hepatic expression levels of the cytochrome P450 (CYP), regulate the hepatic clearance of Clz, thereby determine its bioavailability.

The CYP1A2 and CYP2C19 isoenzymes are mainly responsible for the metabolism of several drugs including Clz. It has been demonstrated that there is an interethnic variation in the expression and function of these two isoenzymes. This variation is caused by single nucleotide polymorphisms (SNPs) of genes encoding these proteins.

While the Influence of the different polymorphisms related to CYP1A2 and CYP2C19 have been established especially in Asian and Caucasian populations, no study has examined the impact of these SNPs in the southern Mediterranean populations. Moreover, the impact of these SNPs is very controversial. The present study aims to investigate in Tunisian schizophrenic patients, the influence of genetic (CYP1A2 and CYP2C19 polymorphisms) and non-genetic factors on Clz pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenic patients receiving clozapine
* Good adherence to the treatment (clozapine)

Exclusion Criteria:

* Patients who were co-prescribed drugs that affected the pharmacokinetics of Clozapine.
* Patients who presented gastrointestinal disorders disturbing absorption of clozapine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2019-12-14 (Actual)

PRIMARY OUTCOMES:
Determination of trough plasma concentration of clozapine (C0) | One and a half months
  Technique : HPLC/UV (high-performance liquid chromatography associated with a UV detector)

SECONDARY OUTCOMES:
Determination of the correlation between the presence of CYP1A2*1F (rs762551;-163C> A), CYP1A2*1C (rs2069514;-3860 G> A) and CYP 2C19*2 (rs4244285; 681G>A) and the variability of C0/Daily dose. | One and a half months
  - Technique: PCR-RFLP (Polymerase Chain Reaction-Restriction Fragment Length Polymorphism)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medecine of Monastir, Monastir, Tunisia